CLINICAL TRIAL: NCT01342497
Title: A Randomised, Double-Blind, Repeat-Dose, Placebo-Controlled Phase IIa Proof of Concept Study to Investigate the Safety and Efficacy of Oral BBR-012 in Combination With Standard Medical Care in Diabetic Patients With Complicated Skin Ulceration on the Foot (Diabetic Foot Ulcer)
Brief Title: Oral BBR-012 in the Treatment of Diabetic Foot Ulcers, Proof of Concept Study
Acronym: BBR-012
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bridge BioResearch Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBR-012CS01
Record Dates: First submitted 2011-04-12; First posted 2011-04-27 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BBR-012 (Experimental)
  Interventions: Drug: isoniazide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: isoniazide — Tablets, dosing 3 times daily, 12 weeks
  Arms: BBR-012
Drug: placebo — tablets, dosing 3 times daily, 12 weeks
  Arms: Placebo

SUMMARY:
The aim of this Clinical Proof of Principle study is to evaluate the effect of BBR-012 on the healing of complicated diabetic foot ulcers.

ELIGIBILITY:
Main Inclusion Criteria:

* Aged ≥18
* Diabetes mellitus
* Ischaemic or neuro-ischaemic Diabetic Foot Ulcer below the malleolus, but not wholly on the sole of the foot (minimum size: 1 cm x 1 cm)
* Body Mass Index(BMI) ≤40 kg/m2
* Women of childbearing potential must use acceptable methods of birth control
* Written informed consent to participate in the study
* Patients must be able to speak English fluently and to understand English

Main Exclusion Criteria:

* Any uncontrolled illnesses (e.g. active malignancy, vasculitis) that, in the opinion of the investigator, would interfere with interpreting the results of the study
* Infected Diabetic Foot Ulcer based on the IDSA guidelines, i.e. presence of purulent secretions or at least two of the manifestations of inflammation (erythema, warmth, swelling or induration and pain or tenderness), and for whom, in the investigator's judgment, intravenous or oral antibiotic therapy is required
* Active osteomyelitis
* Wholly plantar Diabetic Foot Ulcer
* Suspected gangrenous tissue of the affected limb that cannot be removed with a single debridement
* Diabetic Foot Ulcer associated with prosthetic material or a device
* Received any potentially effective systemic antibiotic therapy for more than 24 hours during the 72-hour period before the screening visit
* Is receiving, or has received within the 14 days prior to the screening visit, any concomitant topical wound therapy (e.g., topical antimicrobial therapy, topical debriding agent, topical growth factor, topical skin replacement, or hyperbaric oxygen)
* Has received systemic corticosteroids, immunosuppressive agents, radiation therapy or chemotherapy within the 30 days prior to the screening visit.
* Hepatic impairment, renal impairment (defined as estimated glomerular filtration rate <10 mL/minute/1.73m2), hypersensitivity to isoniazid.
* High risk for tuberculosis, e.g. HIV positive, are immunosuppressed, or have active malignancy
* Symptoms of active or latent tuberculosis (based on specific history, physical examination, Interferon Gamma Release Assay (IGRA) test and chest X-Ray)
* Known or suspected drug or alcohol abuse or positive drugs of abuse test.
* Participating in any clinical study the 12 weeks before the screening visit
* Donation of more than 450 mL of blood in the 3 months before the screening visit, or 1200 mL blood in the 12 months before the screening visit.
* History of severe hypersensitivity or ongoing hypersensitivity that might affect the patient's suitability for the study (e.g. hypersensitivity to wound dressings), as judged by the investigator.
* History of allergy to, or insensitivity to, local anaesthetics
* Use of any prescribed or non-prescribed (over-the-counter) medication, including herbal medication (e.g., St. Johns Wort) that could possibly interfere with the objectives of this study (e.g., could affect the closure of chronic dermal ulceration), during 2 weeks (or 5 half-lives of the compound whichever is the longer) before the anticipated first dose of study medication. Occasional paracetamol for pain relief (maximum 2 g per 24 hours) and adrenergic nasal spray for relief of nasal congestion are allowed
* Having received BBR-012 or isoniazid within the 6 months prior to the screening visit
* Bleeding disorder or history of increased bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Rate of healing of diabetic foot ulcers (% reduction in area from baseline) | 4, 8 and 12 weeks

SECONDARY OUTCOMES:
Rate of healing (change from baseline) as assessed by various scoring criteria: IDSA, modified ASEPSIS score, TEXAS Diabetic wound score, composite severity score and global clinical assessment | week 1, 2, 3, 4, 6, 8, 10, 12 and 13-14(follow up)
Effect of BBR-012 on the level of ischemia (change from baseline as measured by tcpO2) | 4, 8 and 12 weeks
Effect of BBR-012 on microbiological outcome (presence of pathogens and outcome as compared to baseline) | week 1, 2, 3, 4, 6, 8, 10, 12 and 13-14(follow up)
Safety and tolerability of BBR-012 as assessed by reported adverse events and safety laboratory parameters | from baseline visit to week 14

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Boulton, Professor, Principal Investigator — Manchester Royal Infirmary
Locations (11):
- United Kingdom (11):
  - Tameside Hospital NHS Foundation Trust, Ashton-under-Lyne
  - Bradford Royal Infirmary , Bradford Teaching Hospitals NHS Trust, Bradford
  - Department of Wound Healing, School of Medicine, Cardiff University, Cardiff
  - Chorley & South Ribble Hospital, Lancashire Teaching Hospitals Trust, Chorley
  - Croydon University Hospital, Croydon
  - Royal Infirmary of Edinburgh, Lothian University Hospital Trust, Edinburgh
  - Gloucester Royal Hospital NHS Foundation Trust, Gloucester
  - Manchester Royal Infirmary, University Department of Medicine, Manchester
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth Hospitals NHS Trust, Plymouth
  - Southampton Hospitals NHS Trust, Southampton